CLINICAL TRIAL: NCT07157267
Title: Evaluation of Thyroid Function, Lipid Profile, and Uric Acid Levels in Patients Undergoing Hemodialysis Prevalence in Assiut University Hospital
Brief Title: Evaluation of Thyroid Function, Lipid Profile, and Uric Acid Levels in Hemodialysis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nermen Maher, resident at the Internal Medicine Department, Assiut University
Other Study IDs: Hemodialysis Patients
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Dysfunction; Hemodialysis; Elevated Uric Acid
Keywords: hemodialysis; elevated uric acid; Thyroid Function Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population consists of adult patients aged 18 years or older, undergoing regular hemodialy: The study involves 100 adult patients (≥18 years) who are on maintenance hemodialysis for three months or more. Patients with any known thyroid disorder prior to starting dialysis, those receiving lipid-lowering agents or uric acid-lowering medications, and those recently hospitalized or with acute infections in the last month are excluded. The population reflects a typical CKD hemodialysis demographic seen at Assiut University Hospital and includes diverse participants with varying ages, genders, smoking histories, and comorbid conditions such as diabetes mellitus and hypertension. Clinical and demographic data will be systematically gathered, including dialysis durations and adequacy, to provide comprehensive insights into the interplay of thyroid, lipid, and uric acid metabolism in these patients.

SUMMARY:
This observational study evaluates the prevalence and relationships of thyroid dysfunction, lipid abnormalities, and elevated uric acid levels in adult patients undergoing maintenance hemodialysis at Assiut University Hospital.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) patients on maintenance hemodialysis frequently experience metabolic disturbances including thyroid hormone imbalances, dyslipidemia, and hyperuricemia, which heighten cardiovascular risk. This prospective cross-sectional study aims to investigate the prevalence and interrelations of thyroid function abnormalities (measured via serum TSH, Free T3, Free T4), lipid disorders (total cholesterol, HDL-C, LDL-C, triglycerides), and serum uric acid levels in a cohort of 100 adult patients undergoing regular hemodialysis for at least three months at Assiut University Hospital. Data will be collected through questionnaires, clinical exams, ultrasound thyroid scanning, and detailed laboratory and dialysis records review. The study also examines correlations between these biochemical parameters and patients' demographic and clinical characteristics, such as age, gender, smoking status, dialysis duration/frequency, and comorbidities like diabetes mellitus and hypertension. Statistical analyses using SPSS will identify the prevalence of metabolic alterations and their clinical implications in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* On regular hemodialysis for ≥3 months

Exclusion Criteria:

* On lipid-lowering or uric acid-lowering medications
* Acute infections or hospitalizations in the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study population consists of adult patients aged 18 years or older, undergoing regular hemodialysis treatment at Assiut University Hospital for a minimum of three months, excluding those with pre-existing thyroid disorders or on relevant medications.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Thyroid Function Status | baseline
  Assessment of the prevalence and types of thyroid dysfunction in hemodialysis patients

REFERENCES:
- [Background] Liu WC, Tomino Y, Lu KC. Impacts of uric acid on chronic kidney disease progression: a review. J Adv Res. 2017;8(5):449-56.